CLINICAL TRIAL: NCT04115228
Title: Clinical Feasibility Study, Implantable Tibial Nerve Stimulator (ITNS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nine Continents Medical, Inc. (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ITNS-01; R44DK121578 (NIH)
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-03

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Study device (Experimental): Subjects who provide informed consent, meet all inclusion criteria, and no exclusion criterion, will have a study device implanted and followed closely for 26 weeks.
  Interventions: Device: Implantation and neuromodulation therapy

INTERVENTIONS:
Device: Implantation and neuromodulation therapy — The study device is an autonomous permanent implant for neuromodulation targeting the posterior tibial nerve. It does not require an external power source or charger.
  Other Names: Nine Continents Medical ITNS model 9C-680

SUMMARY:
Study objectives: To report feasibility data for safety and effectiveness of the study device.

Study device: Nine Continents Medical implantable tibial nerve stimulator (ITNS) model 9C-680 with programmer model 9C-580.

Intended use: The study device is intended for treatment of the symptoms of overactive bladder (OAB), including urinary urge incontinence and significant symptoms of urgency-frequency alone or in combination, in patients who have failed or could not tolerate more conservative treatments.

Type of design: Single-arm longitudinal design.

Study sites: Single site, in the United States.

Study duration: One year total, comprising six months for enrolling and implanting 10 subjects, and 26 weeks for follow-up.

ELIGIBILITY:
Inclusion Criteria:

At pre-screening:

* Age 18 years or older;
* Documented diagnosis of overactive bladder;
* Documented failed behavioral intervention and/or physical therapy;
* Documented failed first drug for overactive bladder; and
* Documented failed second drug for overactive bladder.

At screening:

* Life expectancy of at least one year;
* Capable of tolerating the implantation procedure;
* Ambulatory and able to use the toilet independently and without difficulty; and
* Able to sense and tolerate posterior tibial nerve stimulation (transcutaneous test).

Based on pre-therapy voiding diary:

* Average daily voids during waking hours ≥ 11;
* Average daily voids interrupting sleep ≥ 2.0;
* Average daily voids associated with urgency ≥ 4; or
* Average daily incontinence episodes ≥ 1.

Exclusion Criteria:

At pre-screening:

* Predominant stress incontinence;
* For females, pelvic organ prolapse quantification (POP-Q) ≥ grade II;
* Neurologic disease, e.g. MS, Parkinson's;
* Abnormal upper urinary tract function;
* Neurogenic bladder;
* Bladder stone or tumor;
* Body mass index (BMI) > 40;
* Chronic pelvic pain;
* Urinary fistula;
* Peripheral neuropathy;
* History of failed neuromodulation for overactive bladder;
* Uncontrolled bleeding disorder;
* End stage renal failure, glomerular filtration rate (GFR) < 35, or dialysis;
* Untreated diabetes or A1C > 7;
* Implanted pacemaker, defibrillator, or neurostimulator;
* History of pelvic cancer within the past two years;
* Condition requiring magnetic resonance imaging (MRI);
* Condition requiring diathermy;
* Metallic implant in planned site of study device;
* For females, pregnant;
* For females, planning to become pregnant;
* For females, given birth in the last 6 months; or
* For females, of child-bearing potential and not willing to practice a medically-approved method of birth control during the study.

At screening:

* Anatomical restriction preventing device placement;
* Skin lesions or compromised skin at the implant site;
* For females, pelvic organ prolapse quantification (POP-Q) ≥ grade II;
* Post-void residual > 150 cc;
* Urinary tract mechanical obstruction due to urethral stricture;
* Urinary tract mechanical obstruction due to bladder neck contracture;
* In males, urinary tract mechanical obstruction due to benign prostatic hyperplasia (BPH);
* Vesicoureteral reflux;
* Cystoscopic abnormalities that could be malignant;
* Current cystitis;
* Current urethritis;
* Gross hematuria;
* In females, positive pregnancy test;
* Any other medical condition with potential effect on bladder function, as assessed by investigator; or
* Any other medical condition that could compromise the safety of the subject, as assessed by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parminder Sethi, M.D., Principal Investigator — Pacific Urology
Locations (1):
- Pacific Urology, San Ramon, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sethi PS, Peters KM. A First-In-Human Feasibility Study of a New Implantable Tibial Nerve Stimulator for Overactive Bladder Syndrome. Neuromodulation. 2025 Jul;28(5):832-839. doi: 10.1016/j.neurom.2025.01.013. Epub 2025 Mar 1. PMID 40029222

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Device
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Device
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Met inclusion criterion for incontinence, based on pre-therapy diary [Count of Participants; unit: Participants] | 7
Met inclusion criterion for frequency, based on pre-therapy diary [Count of Participants; unit: Participants] | 2
Met inclusion criterion for nocturia, based on pre-therapy diary [Count of Participants; unit: Participants] | 7
Met inclusion criterion for urgency, based on pre-therapy diary [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Urinary Incontinence Frequency From Baseline to 13 Weeks
Description: For a participant analyzed, let x0 = average number of voids with leakage per 24 hours in first 72 hours of baseline diary, x1 = average number of voids with leakage per 24 hours in first 72 hours of 13-week diary, and x = percent change of urinary incontinence frequency from baseline to 13 weeks.
  Then x = 100 * (x1 - x0) / x0. For example, a participant with an average of 4 voids with leakage per 24 hours in the first 72 hours of the baseline diary and 2 voids with leakage per 24 hours in the first 72 hours of the 13-week diary would have a percent change of urinary incontinence frequency from baseline to 13 weeks of 100 * (2 - 4) / 4 = -50.
Time Frame: Baseline to 13 weeks
Population: Subjects who met the inclusion criterion for incontinence
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Study Device
Number analyzed (Participants) | 7
percent change | -89 (14)

2. Primary Outcome: Percent Change of Excess Voiding Frequency During Waking Hours From Baseline to 13 Weeks
Description: For a participant analyzed, let x0 = average number of voids during waking hours per 24 hours in first 72 hours of baseline diary, x1 = average number of voids during waking hours per 24 hours in first 72 hours of 13-week diary, and x = percent change of excess voiding frequency during waking hours from baseline to 13 weeks, where "excess" means voids during waking hours exceeding 7 per 24 hours.
  Then x = 100 * (x1 - x0) / (x0 - 7). For example, a participant with an average of 16 voids during waking hours per 24 hours in the first 72 hours of the baseline diary and an average of 10 voids during waking hours per 24 hours during the first 72 hours of the 13-week diary would have a percent change of excess voiding frequency during waking hours from baseline to 13 weeks of 100 * (10 - 16) / (16 - 7) = -67.
Time Frame: Baseline to 13 weeks
Population: Subjects meeting inclusion criterion for frequency at baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Study Device
Number analyzed (Participants) | 2
percent change | -90 (33)

3. Primary Outcome: Percent Change of Frequency of Voids Awakening From Sleep From Baseline to 13 Weeks
Description: For a participant analyzed, let x0 = average number of voids awakening from sleep per 24 hours in first 72 hours of baseline diary, x1 = average number of voids awakening from sleep per 24 hours in first 72 hours of 13-week diary, and x = percent change of frequency of voids awakening from sleep from baseline to 13 weeks.
  Then x = 100 * (x1 - x0) / x0. For example, a participant with an average of 2 voids awakening from sleep per 24 hours in the first 72 hours of the baseline diary and an average of 1 void awakening from sleep per 24 hours during the first 72 hours of the 13-week diary would have a percent change of frequency of voids awakening from sleep from baseline to 13 weeks of 100 * (1 - 2) / 2 = -50.
Time Frame: Baseline to 13 weeks
Population: Subjects meeting inclusion criterion for nocturia at baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Study Device
Number analyzed (Participants) | 7
percent change | -30 (25)

4. Primary Outcome: Percent Change of Frequency of Voids With Urgency From Baseline to 13 Weeks
Description: For a participant analyzed, let x0 = average number of voids with urgency per 24 hours in first 72 hours of baseline diary, x1 = average number of voids with urgency per 24 hours in first 72 hours of 13-week diary, and x = percent change of frequency of voids with urgency from baseline to 13 weeks, where "voids with urgency" means voids self-reported with some or severe urgency, or leakage.
  Then x = 100 * (x1 - x0) / x0. For example, a participant with an average of 8 voids with urgency per 24 hours in the first 72 hours of the baseline diary and an average of 5 voids with urgency per 24 hours during the first 72 hours of the 13-week diary would have a percent change of frequency of voids with urgency from baseline to 13 weeks of 100 * (5 - 8) / 8 = -37.5
Time Frame: Baseline to 13 weeks
Population: Subjects meeting inclusion criterion for urgency at baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Study Device
Number analyzed (Participants) | 10
percent change | -69 (23)

5. Secondary Outcome: Threshold at 13 Weeks
Description: Neuromodulation pulse amplitude required to evoke paresthesia or motor response ("threshold") at 13 weeks.
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | Study Device
Number analyzed (Participants) | 10
Volts | 1.03 (0.94)

6. Secondary Outcome: Change of Score on an Overactive Bladder Questionnaire Short-form (OAB-q SF) Symptom Bother Subscale From Baseline to 13 Weeks
Description: The overactive bladder questionnaire short-form (OAB-q SF) symptom bother subscale ranges from 0 to 100, and higher symptom bother scores indicate greater symptom bother ( worse outcome).
  For a participant analyzed, let x0 = symptom bother score at baseline, x1 = symptom bother score at 13 weeks, and x = x0 - x1. For example, a participant with a symptom bother score of 60 at baseline and a symptom bother score of 20 at 13 weeks would have a change of score on the overactive bladder questionnaire short-form (OAB-q SF) symptom bother subscale from baseline to 13 weeks of -40.
Time Frame: Baseline to 13 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Study Device
Number analyzed (Participants) | 10
Scores on a scale | -40 (16)

7. Secondary Outcome: Score on a Global Response Assessment (GRA) Scale at 13 Weeks
Description: The global response assessment (GRA) scale ranges from 1 to 6, with 1 corresponding to "markedly worse" and 6 corresponding to "markedly better", so that higher scores represent better outcomes..
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Study Device
Number analyzed (Participants) | 10
Score on a scale | 5.8 (0.4)

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Study Device
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Device (N=10)
Incision-site issue (Skin and subcutaneous tissue disorders) | 4 (10) — Three (3) subjects experienced redness at the site (cause undetermined) and of these, 2 resolved with treatment, and 1 resolved spontaneously. One (1) had a positive bacterial culture at the site, which resolved with treatment.
Urinary tract infection (Renal and urinary disorders) | 2 (10) — Not device or procedure related.
Previously-planned surgery for unrelated issue (Surgical and medical procedures) | 2 (10) — One (1) subject had surgery for torn tendon and/or ligaments in right shoulder. One (1) had total replacement of right knee.
Unconfirmed report that implant "stopped working" (Product Issues) | 1 (10) — Subject's impression could not be confirmed. Device check showed normal operation. Subject completed a voiding diary at 13 weeks, which showed responder status.

LIMITATIONS AND CAVEATS:
Clinical feasibility study with single-arm design, single investigator, and small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For this clinical feasibility study, the investigator agrees to maintain confidentiality and refrain from publication without the sponsor's prior written approval.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT04115228/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT04115228/ICF_001.pdf